CLINICAL TRIAL: NCT03071913
Title: Pilot Study to Assess Heterogeneity of the Blood Brain Barrier in Patients with CNS Malignancy
Brief Title: Blood Brain Barrier Differences in Patients with Brain Tumors Undergoing Surgery
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: MC1671; U54CA210180 (NIH); NCI-2017-00299 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16-007782 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2017-02-27; First posted 2017-03-07 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-04

CONDITIONS: Central Nervous System Neoplasm; Localized Brain Neoplasm; Metastatic Malignant Neoplasm in the Brain; Recurrent Brain Neoplasm
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (biospecimen collection): As part of pre-operative standard of care, patients receive levetiracetam by injection and cefazolin by injection. Patients are also offered lorazepam in the pre-operative area. At the time of surgery, patients undergo approximately 2 tissue biopsies from 3-4 tumor locations. This tissue is removed as part of the planned surgery, but it is also tested for research purposes. During surgery, a blood sample is collected every 20-30 minutes beginning at the time of skin incision until all of the research tumor samples have been removed. A minimum of 3 blood samples are collected up to a maximum of 12.
  Interventions: Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of tissue and blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot research trial studies blood brain barrier differences in patients with brain tumors undergoing surgery. Studying samples of tissue and blood from patients with brain tumors in the laboratory may help doctors to understand how well drugs get into different parts of a brain tumor. This may help them to determine which types of drugs may be best for treating brain tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To define the heterogeneity of blood brain barrier (BBB) permeability by assessing drug distribution in a population of patients with central nervous system (CNS) malignancy.

SECONDARY OBJECTIVE:

I. Establish correlation of BBB permeability with radiographic appearance for study patients.

CORRELATIVE RESEARCH OBJECTIVE:

I. To utilize tumor samples to investigate mechanisms for BBB heterogeneity.

OUTLINE:

As part of pre-operative standard of care, patients receive levetiracetam by injection and cefazolin by injection. Patients are also offered lorazepam in the pre-operative area. At the time of surgery, patients undergo approximately 2 tissue biopsies from 3-4 tumor locations. This tissue is removed as part of the planned surgery, but it is also tested for research purposes. During surgery, a blood sample is collected every 20-30 minutes beginning at the time of skin incision until all of the research tumor samples have been removed. A minimum of 3 blood samples are collected up to a maximum of 12.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Clinical and radiographic evidence suggesting CNS malignancy
* Suspected newly diagnosed, local, or intracranial recurrence of primary brain tumor OR previously untreated or treated brain metastasis
* Willing to undergo a neurosurgical resection of CNS lesion at Mayo Clinic Rochester
* Able to have magnetic resonance imaging (MRI) imaging with gadolinium contrast (e.g. no cardiac pacemaker, defibrillator, renal failure)
* Females of childbearing potential must have a negative pregnancy test done =< 14 days prior to registration
* Provide written informed consent
* Willing to provide tissue and blood samples for research purposes
* Patients having a study-specific surgical planning MRI only: Creatinine (estimated glomerular filtration rate [eGFR] >= 30) (obtained =< 30 days prior to registration)

Exclusion Criteria:

* Vulnerable populations: pregnant women, prisoners, mentally handicapped
* Unable to undergo a biopsy of CNS lesion
* Documented drug allergy to cefazolin or levetiracetam, or other contraindication to use these drugs in the pre-operative setting (e.g., patient is already on another anti-seizure medication which precludes the clinical indication for pre-operative levetiracetam)
* Patients who are unable to swallow tablets if study drug is administered by mouth
* Patients who are at risk for impaired absorption of oral medication if study drug is administered by mouth; Note: This includes but not limited to, refractory vomiting, gastric resection/bypass, and duodenal/jejunal resection
* Pregnant or nursing women; Note: Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects with chemotherapy; there is also a potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with these drugs, so breastfeeding should be discontinued for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CNS malignancy
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Blood brain barrier permeability as measured by the ratio of drugs in blood and tissue samples taken during surgery | At the time of surgery
  The ratio of cefazolin and levetiracetam (or lorazepam) and gadolinium in blood taken every 20-30 minutes during surgery will be correlated with the tissue samples. Inter- and intra-subject variability over all patients will be estimated, within specific imaging features between patients, and within open biopsy specimens.

SECONDARY OUTCOMES:
Radiographic appearance at each tissue sample location | At the time of surgery
  The results of the tissue samples will be compared with the radiographic appearance at each tissue sample location. This will be primarily descriptive in nature.

CONTACTS AND LOCATIONS:
Overall Officials: Jann N. Sarkaria, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials